CLINICAL TRIAL: NCT01203189
Title: Seborrheic Dermatitis of the Scalp in Populations Practicing Less Frequent Hair Washing: Ketoconazole 2% Foam Versus Ketoconazole 2% Shampoo
Brief Title: Seborrheic Dermatitis: Ketoconazole 2% Foam Versus Ketoconazole 2% Shampoo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Aibing M. Guo, MD, Assistant Professor, St. Louis University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: seb derm 2010
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Seborrheic Dermatitis
Keywords: dandruff, flaky scalp
MeSH Terms: conditions — Dermatitis, Seborrheic; Dandruff | interventions — Ketoconazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Shampoo Group (Active Comparator): Subjects in the S group will wash their hair twice weekly for four weeks with ketoconazole 2% shampoo.
  Interventions: Drug: ketoconazole 2% shampoo
- Foam group (Active Comparator): Subjects in the F group will apply ketoconazole 2% foam to the scalp twice daily for four weeks.
  Interventions: Drug: ketoconazole 2% foam
- Cross Over Group (Active Comparator): apply ketoconazole 2% foam to scalp twice daily for four weeks. Subjects in the Shampoo group will be able to cross over into the Foam group if the TDSS score does not improve by 60% at the end of the four week treatment period using shampoo.
  Interventions: Drug: ketoconazole 2% foam; Drug: ketoconazole 2% shampoo

INTERVENTIONS:
Drug: ketoconazole 2% foam — Subjects in the Foam (F) group will apply ketoconazole 2% foam to the scalp twice daily for four weeks.
  Other Names: Extina
  Arms: Cross Over Group; Foam group
Drug: ketoconazole 2% shampoo — Subjects in the Shampoo (S) group will wash their hair twice weekly for four weeks with ketoconazole 2% shampoo.
  Other Names: Nizoral
  Arms: Cross Over Group; Shampoo Group

SUMMARY:
The aims of this study are to compare the effectiveness of antifungal foam versus antifungal shampoo and determine patient compliance and satisfaction with both vehicles among African American females with dandruff practicing less than once weekly hair washing.

DETAILED DESCRIPTION:
A wide variety of topical vehicles are available for medications that treat scalp disorders. Proper vehicle selection is important when managing scalp conditions, such as seborrheic dermatitis, because the efficacy of these treatments depends largely on compliance and the amount of active ingredient delivered to the scalp. It is therefore important to prescribe vehicles that are easy to apply and cause the least amount of disruption to the patients' pre-existing hair care practices. One of the most common rate limiting hair care practices among different cultures is wash frequency. Literature shows African American women are more likely to wash their hair less than once weekly versus Caucasian women. We hypothesize certain vehicles, such as foam preparations which do not require hair washing, will be more efficacious in African American women with seborrheic dermatitis than shampoo preparations.

ELIGIBILITY:
Inclusion Criteria:

* African American females aged 18 to 89 years
* Previous diagnosis of seborrheic dermatitis of the scalp
* TDSS between 50 and 200
* Practice less than or equal to once weekly hair washing
* Immunocompetent
* Willing to not grease or oil scalp

Exclusion Criteria:

* Age below 18 years or above 89 years
* Medical history of psoriasis, diabetes mellitus, immunosuppression, neurologic disorders, and/or chronic disease not stabilized by medication
* Patients taking any oral steroids and/or antifungals within 30 days of enrollment
* Sensitivity to any formulation components of either ketoconazole foam or shampoo including sulfur
* The use of any topical medications including over the counter products indicated for the treatment of seborrheic dermatitis within 14 days of enrollment
* Pregnant women, women who plan on becoming pregnant, or breastfeeding women
* Current use or history of using any biologic medication

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aibing M Guo, M.D., Principal Investigator — St. Louis University Dermatology; Scott W Fosko, M.D., Study Chair — St. Louis University Dermatology
Locations (1):
- St. Louis University Department of Dermatology, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Shampoo Only Group: Subjects in the S group will wash their hair twice weekly for four weeks with ketoconazole 2% shampoo.
  ketoconazole 2% shampoo: Subjects in the S group will wash their hair twice weekly for four weeks with ketoconazole 2% shampoo.
- Foam Only Group: Subjects in the F group will apply ketoconazole 2% foam to the scalp twice daily for four weeks.
  ketoconazole 2% foam: Subjects in the F group will apply ketoconazole 2% foam to the scalp twice daily for four weeks.
- Shampoo First and Then Foam: subjects used shampoo for 4 weeks, but did not reach 60% improvement on TDSS score were given foam treatment for 4 weeks
Period: First 4 Weeks Treatment
Arm/Group | Shampoo Only Group | Foam Only Group | Shampoo First and Then Foam
Started | 10 | 10 | 3
Completed | 8 | 8 | 3
Not Completed | 2 | 2 | 0
Period: Cross Over Period 4 Weeks Treatment
Arm/Group | Shampoo Only Group | Foam Only Group | Shampoo First and Then Foam
Started | 0 | 0 | 3
Completed | 0 | 0 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects in the S group were able to cross over into the F group if the TDSS score does not improve by 60% at the end of the 4 week treatment period. These cross over subjects remained in the study for an additional 4 weeks to apply ketoconazole foam 2%. The 4 subject in the cross over group were originally in the shampoo group.
Groups:
- Shampoo Group: Subjects in the S group will wash their hair twice weekly for four weeks with ketoconazole 2% shampoo.
  ketoconazole 2% shampoo: Subjects in the S group will wash their hair twice weekly for four weeks with ketoconazole 2% shampoo.
- Foam Group: Subjects in the F group will apply ketoconazole 2% foam to the scalp twice daily for four weeks.
  ketoconazole 2% foam: Subjects in the F group will apply ketoconazole 2% foam to the scalp twice daily for four weeks.
- Cross Over Group: Subjects in the Shampoo group will be able to cross over into the Foam group if the TDSS score does not improve by 60% at the end of the four week treatment period. These cross over subjects will remain in the study for an additional four weeks and apply foam in the same manner as subjects in the original Foam group.
  ketoconazole 2% foam: Subjects in the F group will apply ketoconazole 2% foam to the scalp twice daily for four weeks.
- Total: Total of all reporting groups
Arm/Group | Shampoo Group | Foam Group | Cross Over Group | Total
Number analyzed (Participants) | 10 | 10 | 3 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 3 | 23
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 3 | 23
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 3 | 23

OUTCOME MEASURES:

1. Primary Outcome: Total Dandruff Severity Score (TDSS)
Description: The scalp will be divided into quadrants and for each quadrant the percent of involvement and degree of severity will be assessed. The percent of involvement will be measured on a scale of 0 to 4 in which a score of 0 means less than 10% involvement, and a score of 4, more than 76% involvement. Severity will be measured on a scale of 0 to 3 in which a score of 0 indicates normal skin, and a score of 3, marked erythema with thick confluent plates of yellowish white scales. The whole scalp score will then calculated by multiplying the total percent involvement score by the total severity score.
  Quadrant scalp score = percent involvement score x severity score Total scalp score = summation of all the quadrant scores TDSS value ranges from 0-48, with 0 equal to no scale, which is the best outcome, compared to 48, which is the most severe and worse outcome
Time Frame: up to 8 weeks
Population: Data were not collected for the Shampoo only group and Foam Only group at 8 weeks. Only 3 participants completed the 8 weeks of cross over treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Shampoo Only Group | Foam Only Group | Cross Over Group
Number analyzed (Participants) | 8 | 8 | 3
units on a scale
  Baseline TDSS score | 28.6 (11.0) | 29.3 (13.2) | 26.7 (16.2)
  TDSS at 4 weeks | 2.1 (3.8) | 5.6 (7.1) | 33.7 (19.9)
  TDSS at 8 weeks: number analyzed (Participants) | 0 | 0 | 3
  TDSS at 8 weeks |  |  | 8.7 (0.6)

2. Secondary Outcome: Number of Participants Who Are Always Compliant.
Description: Patient compliance will be evaluated by having patients keep a diary documenting the use of study drug. They will also be questioned about their medication usage at every visit. In addition, we will weigh the study drug at every visit.
  a patient is classified as always indicates that they use their medicine as directed on their diary on every visit.
Time Frame: at end of each treatment period (4 weeks and 8 weeks)
Population: Data were not collected for the Shampoo Only Group and Foam Only Group at end of 8 weeks. Only 3 participants finished the study in the Cross Over Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Shampoo Only Group | Foam Only Group | Cross Over Group
Number analyzed (Participants) | 8 | 8 | 3
Participants
  compliance at week 4 | 7 | 3 | 1
  compliance at week 8: number analyzed (Participants) | 0 | 0 | 3
  compliance at week 8 |  |  | 0

3. Secondary Outcome: Number of Participants Who Are Very Satisfied
Description: Patient satisfaction will be measured using a five point satisfaction scale.
  1. very dissatisfied
  2. dissatisfied
  3. Neutral
  4. satisfied
  5. very satisfied.
Time Frame: data were collected at end of each treatment period (4 weeks and 8 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Shampoo Only Group | Foam Only Group | Cross Over Group
Number analyzed (Participants) | 8 | 8 | 3
Participants
  Very Satisfied at 4 weeks | 5 | 8 | 0
  Very Satisfied at 8 weeks: number analyzed (Participants) | 0 | 0 | 3
  Very Satisfied at 8 weeks |  |  | 0

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Shampoo Only Group | Foam Only Group | Cross Over Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/3
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/3

LIMITATIONS AND CAVEATS:
1. Small Sample Size.
2. Unable to control for wash frequency between the two groups, i.e. shampoo group vs foam group.
3. Study group was comprised of patients with moderate seborrheic dermatitis, results may vary in mild or severe cases.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No